CLINICAL TRIAL: NCT04417543
Title: Effect of Memantine on Cognitive Impairment in Patients With Epilepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Mohmed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Memantine in epilepsy
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: 100 patients divided into two groups each group 50patients
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Memantine hydrochloride group (Active Comparator): included 50 patients who received memantine
  Interventions: Drug: Memantine Hydrochloride
- Placebo group (Placebo Comparator): included 50 patients who received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine Hydrochloride — Memantine is a low-affinity voltage-dependent uncompetitive antagonist of the NMDA-type glutamate receptor .Memantine hydrochloride tablet was started at the dose of 5 mg once daily orally, and the same dose was given for 3months and dose is titrated to 10 mg once daily orally for the remaining 3months. Placebo was given once daily orally for6months. Patients were instructed to take the study medication at the same time every day.
  Other Names: Memantine
  Arms: Memantine hydrochloride group
Drug: Placebo — Placebo was given once daily orally for6months. Patients were instructed to take the study medication at the same time every day.
  Arms: Placebo group

SUMMARY:
Evaluate the efficacy of memantine on improving the cognitive impairment in patient with epilepsy

DETAILED DESCRIPTION:
Epilepsy is a complex disorder, which involves much more than seizures, encompassing a range of associated comorbid health conditions that can have significant health and quality-of-life implications. Of these comorbidities, cognitive impairment is one of the most common and distressing aspects of epilepsy.

Excito-toxicity, mediated by glutamate acting on N-methyl-D-aspartate (NMDA) receptors in the hippocampus, can cause memory dysfunction in epilepsy .

Memantine is a low-affinity voltage-dependent uncompetitive antagonist of the NMDA-type glutamate receptor . It also has antioxidant property and increases production of brain derived neurotropic factor (BDNF)

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic epilepsy.
* Normal brain imaging (CT brain).
* Patients on anti epileptic drugs more than 6 months.
* No more than two fits per month.
* Score of Mini mental state examination (10-24), mild and moderate cognitive impairment.
* No other medical disorders.

Exclusion Criteria:

* Progressive neurological diseases.
* Abnormal brain imaging (CT brain).
* More than two fits per month.
* Patients with severe cognitive impairment, score of MMSE less than10.
* Patients with severe medical disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Memory Assessment Scale (MAS) | 1.5years
  This comprehensive battery assesses short-term, verbal and visual memory functioning.
Wechsler Adult Intelligence Scale (WAIS) | 1.5years
  Intelligence quotient (IQ) tests are the primary clinical instruments used to measure adult and adolescent intellience.
Brief Visuospatial Memory Test-Revised (BVMT-R) | 1.5years
  The current revised version of the BVMT, a visual display of six simple figures arranged in a 2 × 3 matrix on an 8 × 11 booklet is shown to participants for three consecutive 10-second trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Salma Mohmed Fahmy, Asyut, Egypt

REFERENCES:
- [Background] Bell B, Lin JJ, Seidenberg M, Hermann B. The neurobiology of cognitive disorders in temporal lobe epilepsy. Nat Rev Neurol. 2011 Mar;7(3):154-64. doi: 10.1038/nrneurol.2011.3. Epub 2011 Feb 8. PMID 21304484
- [Background] Aggleton JP. Multiple anatomical systems embedded within the primate medial temporal lobe: implications for hippocampal function. Neurosci Biobehav Rev. 2012 Aug;36(7):1579-96. doi: 10.1016/j.neubiorev.2011.09.005. Epub 2011 Sep 24. PMID 21964564
- [Background] Alvarez PS, Simao F, Hemb M, Xavier LL, Nunes ML. Effects of undernourishment, recurrent seizures and enriched environment during early life in hippocampal morphology. Int J Dev Neurosci. 2014 Apr;33:81-7. doi: 10.1016/j.ijdevneu.2013.12.004. Epub 2013 Dec 21. PMID 24365760